CLINICAL TRIAL: NCT05834179
Title: Effect of Colding of Endotracheal Tubes on Postoperative Sore Throat: A Prospective Randomized Study
Brief Title: Effect of Colding of Endotracheal Tubes on Sore Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Sibel Catalca, Principal Investigator, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KA 23-42
Record Dates: First submitted 2023-04-02; First posted 2023-04-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Sore Throat
Keywords: endotracheal tube; sore throat; dysphagia
MeSH Terms: conditions — Pharyngitis; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cold endotracheal tube (ETT) (Experimental): Patients who were intubated with an ETT which kept in the fridge.
  Interventions: Other: cold endotracheal tube
- Endotracheal tube (ETT) in the normal temperature (No Intervention): Patients who were intubated with an ETT which kept in the operation room.

INTERVENTIONS:
Other: cold endotracheal tube — patients who were intubated with an ETT which kept in the fridge.
  Arms: cold endotracheal tube (ETT)

SUMMARY:
Postoperative sore throat (POST) is a common and undesirable postoperative symptom that causes patient dissatisfaction. Cold application is a non-invasive, non-pharmacological, cost-effective and effort-effective therapy for pain management. The aim of this study was to evaluate whether colding of ETT can reduce sore throat, dysphagia and dysphonia after endotracheal intubation.

DETAILED DESCRIPTION:
The incidence of postoperative sore throat (POST) has been reported up to 62% following general anaesthesia.It is an undesirable events experienced by patients after general anaesthesia. Various pharmacological agents have been applied to reduce POST, such as lidocaine, ketamine, magnesium, corticosteroids or non-steroidal anti-inflammatory drugs. However, these agents may have some systemic and local side effects. Therefore, various non-pharmacological applications have been investigated to reduce sore throat. Cold application is a non-invasive, cost-effective and effort-effective therapy for pain management. Although the mechanism is not clearly known, it increases the pain threshold, slows cellular metabolism, causes vasoconstriction, and reduces capillary permeability. Therefore, we hypothesized that colding of endotracheal tube may decrease POST associated with airway inflammation. The aim of this study was to evaluate whether colding of ETT can reduce sore throat, dysphagia and dysphonia after endotracheal intubation. The goal of this study is to identify a simple, safe, and inexpensive perioperative intervention to reduce post operative sore throat. This study is a prospective, randomised study involving 116 subjects and they will assessed on the incidence and severity of sore throat, dysphagia and dysphonia at 1. 4. 12. 24. hours after removal of endotracheal tube. Outcomes from this study can be extended to patients who will be receiving general anaesthesia using a endotracheal tube to reduce the incidence and severity of sore throat.

ELIGIBILITY:
Inclusion Criteria:

Patients who were entubated with an ETT. Those who accept the research Elective surgery Patients in American Society of Anaesthesiologists (ASA) I and II class 18 years and over Mallampati classification I and II Operation time more than 1 hour

Exclusion Criteria:

Patients with sore throat and lower respiratory tract infection Patients with a history of allergies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
the incidence of sore throat 1 hour after extubation. | 1 hour after extubation
  Presence of sore throat defined as constant pain, independent of swallowing (0=no. 1=yes)

SECONDARY OUTCOMES:
the severity of sore throat 1 hour after extubation. | 1 hour after extubation
  Severity will be graded by the patient as 0=null; 1=mild; 2=moderate; 3=severe
the incidence of sore throat 4 hour after extubation. | 4 hour after extubation
  Presence of sore throat defined as constant pain, independent of swallowing (0=no. 1=yes)
the severity of sore throat 4 hour after extubation. | 4 hour after extubation
  Severity will be graded by the patient as 0=null; 1=mild; 2=moderate; 3=severe
the incidence of sore throat 12 hour after extubation. | 12 hour after extubation
  Presence of sore throat defined as constant pain, independent of swallowing (0=no. 1=yes)
the severity of sore throat 12 hour after extubation. | 12 hour after extubation
  Severity will be graded by the patient as 0=null; 1=mild; 2=moderate; 3=severe
the incidence of sore throat 24 hour after extubation. | 24 hour after extubation
  Presence of sore throat defined as constant pain, independent of swallowing (0=no. 1=yes)
the severity of sore throat 24 hour after extubation. | 24 hour after extubation
  Severity will be graded by the patient as 0=null; 1=mild; 2=moderate; 3=severe
the incidence of dysphonia | 1 hour after extubation
  Presence of dysphonia defined as difficulty or pain on speaking (0=no. 1=yes)
the incidence of dysphonia | 4 hour after extubation
  Presence of dysphonia defined as difficulty or pain on speaking (0=no. 1=yes)
the incidence of dysphonia | 12 hour after extubation
  Presence of dysphonia defined as difficulty or pain on speaking (0=no. 1=yes)
the incidence of dysphonia | 24 hour after extubation
  Presence of dysphonia defined as difficulty or pain on speaking (0=no. 1=yes)
the incidence of dysphagia | 12 hour after extubation
  Presence of dysphagia defined as difficulty or pain provoked by swallowing
the incidence of dysphagia | 24 hour after extubation
  Presence of dysphagia defined as difficulty or pain provoked by swallowing
the incidence of postoperative respiratory infection | 7 days after operation
  Presence of respiratory infection symptoms such as cough, sputum, rhinorrhea, sore tongue, myalgia or fever

CONTACTS AND LOCATIONS:
Overall Officials: sibel çatalca, dr., Principal Investigator — Baskent University Adana Dr. Turgut Noyan Hospital
Locations (1):
- Baskent University, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu JH, Paik HS, Ryu HG, Lee H. Effects of thermal softening of endotracheal tubes on postoperative sore throat: A randomized double-blinded trial. Acta Anaesthesiol Scand. 2021 Feb;65(2):213-219. doi: 10.1111/aas.13705. Epub 2020 Sep 23. PMID 32926423
- [Background] Kim E, Yang SM, Kwak SG, Park S, Bahk JH, Seo JH. Tracheal tubes lubricated with water to reduce sore throat after intubation: A randomized non-inferiority trial. PLoS One. 2018 Oct 4;13(10):e0204846. doi: 10.1371/journal.pone.0204846. eCollection 2018. PMID 30286145
- See also: article — https://pubmed.ncbi.nlm.nih.gov/32926423/
- See also: article2 — https://pubmed.ncbi.nlm.nih.gov/30286145/